CLINICAL TRIAL: NCT04791631
Title: Does Pre-operative D-chart Score Predict Improvement in VFQ-25 Score Following Surgery for Epiretinal Membrane?
Brief Title: 'Distortion as a Predictor of ERM Surgery Outcome'
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Royal College of Surgeons of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: GN18OP439
Record Dates: First submitted 2021-02-09; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Epiretinal Membrane; Distortion; Quality of Life
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Epiretinal membrane surgery — Surgery for epiretinal membrane i.e. standard 3-port pars plana vitrectomy and epiretinal membrane and internal limiting membrane peel. Phakic patients will undergo cataract surgery.

SUMMARY:
Epiretinal membranes (ERM) consist of an abnormal growth of tissue across the retina and are present about 6% of people aged 50 and over. They can cause symptoms of distortion (straight lines appearing bent) or blurred vision. Management options include observation if asymptomatic, or surgery to peel the membrane if symptomatic. Limited data exists regarding how to identify patients who are most likely to benefit from surgery.

We propose to measure the effects on distortion (using D chart), visual acuity and vision-related quality of life (using a validated vision-related quality of life questionnaire) of ERM surgery. This will allow us to investigate whether pre-operative D chart score can predict subsequent improvement in quality of life following surgery. We hope the results will help patients and VR surgeons decide whether or not to proceed with ERM surgery.

The study will be a prospective case series consisting of patients with symptomatic epiretinal membranes who choose to have epiretinal membrane surgery. The study participants will get standard care with the additional administration of a quality of life questionnaire and measurement of distortion (using a D-chart) at 3 different time points (pre-op, and post-op at 26 and 52 weeks). Recruitment will be in Glasgow, with a possibility of other sites being added on at a later stage.

DETAILED DESCRIPTION:
Epiretinal membranes consist of a proliferation of fibrocellular tissue along the inner aspect of the retina. Over time, this membrane can result in anterior-posterior traction and cause disruption of the retinal architecture, which can lead to symptoms of blurred vision, or distorted vision (with straight lines appearing bent or wavy).

Patients with ERM now constitute one of the most common referrals to the vitreoretinal service. Management of epiretinal membrane includes observation or surgery for severely symptomatic membranes. The surgery consists of vitrectomy and epiretinal +/- inner limiting membrane peel. Currently there is limited evidence to help identify which patients with an epiretinal membrane are the most likely to benefit from this operation, which makes it more difficult for patients to be able to weigh up the benefits and risks of proceeding with this elective procedure.

Our study will measure the effects on distortion (using D chart), visual acuity and quality of life of ERM surgery. Hence it will allow us to investigate whether the pre-op D chart score can predict subsequent improvement in quality of life following surgery. This will provide vitreoretinal surgeons and patients with an evidence base regarding the success of this elective procedure and offer realistic expectations regarding surgical outcomes. Ultimately, we hope that the results of this study will facilitate the decision of whether or not to proceed with ERM surgery.

We plan to recruit patients with an epiretinal membrane who choose to undergo surgery at the time of their clinic appointment within the vitreoretinal service. In addition to standard care, the study participants will undergo measurements of distortion (using a D-chart, duration 5-10 minutes) and fill in a quality of life questionnaire. These measurements will be taken before the operation and at six and twelve months following the operation.

The aims of the study are:

* To investigate the sustained effect of epiretinal membrane surgery on distortion (using D-chart), visual acuity and vision-related quality of life (using NEI VFQ-25 questionnaire)
* To determine the relationship between pre-operative distortion score and post-operative vision-related quality of life score following ERM surgery

Our study will have a larger number of participants with a longer period of follow up (52 weeks) than comparable studies. It will be the first epiretinal membrane study that measures distortion using the D-chart, which we believe to be superior to existing tests (such as the M-chart) which have been used in similar studies.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic epiretinal membrane
2. Patients undergoing vitrectomy and gas surgery, under local or general anaesthetic
3. Able to give informed consent
4. 18 years old and over

Exclusion Criteria:

1. Epiretinal membrane secondary to retinal detachment, uveitis or retinal vascular disease
2. Previous vitreoretinal surgery
3. Pre-existing ophthalmic condition which limits the patient's visual acuity (Documented BCVA 6/36 or worse)
4. Pre-existing ophthalmic conditions which cause metamorphopsia (exudative ARMD, central serous retinopathy)
5. VA < 6/60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epiretinal membranes attending the vitreoretinal clinic at the Tennent Institute of Ophthalmology in Glasgow, UK, and meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
VFQ-25 score at final visit (52 weeks after ERM surgery) | 1 year
  Measure of vision-related quality of life using NEI VFQ-25 quality of life questionnaire, 1 year after surgery for epiretinal membrane

SECONDARY OUTCOMES:
Distortion score pre-operatively and at 26 and 52 weeks after ERM surgery | 1 year
  Distortion score calculated using D-chart
Best-corrected visual acuity pre-operatively and at 26 and 52 weeks after ERM surgery | 1 year
  Visual acuity measured in ETDRS
Vision-related quality of life pre-operatively and at 26 and 52 weeks after ERM surgery | 1 year
  Vision-related quality of life assessed using NEI VFQ-25 quality of life questionnaire
Central retinal thickness pre-operatively and at 26 and 52 weeks after ERM surgery | 1 year
  Central retinal thickness obtained from OCT scans done in clinic

CONTACTS AND LOCATIONS:
Overall Officials: Lona Jawaheer, MBChB, Principal Investigator — NHS Greater Glasgow and Clyde; David Yorston, MBChb, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- NHS Greater Glasgow and Clyde Clinical Research and Development Central Office, Paisley, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dawson SR, Shunmugam M, Williamson TH. Visual acuity outcomes following surgery for idiopathic epiretinal membrane: an analysis of data from 2001 to 2011. Eye (Lond). 2014 Feb;28(2):219-24. doi: 10.1038/eye.2013.253. Epub 2013 Dec 6. PMID 24310238
- [Background] Wong JG, Sachdev N, Beaumont PE, Chang AA. Visual outcomes following vitrectomy and peeling of epiretinal membrane. Clin Exp Ophthalmol. 2005 Aug;33(4):373-8. doi: 10.1111/j.1442-9071.2005.01025.x. PMID 16033349
- [Background] Pournaras CJ, Emarah A, Petropoulos IK. Idiopathic macular epiretinal membrane surgery and ILM peeling: anatomical and functional outcomes. Semin Ophthalmol. 2011 Mar;26(2):42-6. doi: 10.3109/08820538.2010.544237. PMID 21469962
- [Background] Rahman R, Stephenson J. Early surgery for epiretinal membrane preserves more vision for patients. Eye (Lond). 2014 Apr;28(4):410-4. doi: 10.1038/eye.2013.305. Epub 2014 Jan 10. PMID 24406414
- [Background] Ghazi-Nouri SM, Tranos PG, Rubin GS, Adams ZC, Charteris DG. Visual function and quality of life following vitrectomy and epiretinal membrane peel surgery. Br J Ophthalmol. 2006 May;90(5):559-62. doi: 10.1136/bjo.2005.085142. Epub 2006 Jan 18. PMID 16421185
- [Background] Ichikawa Y, Imamura Y, Ishida M. Associations of aniseikonia with metamorphopsia and retinal displacements after epiretinal membrane surgery. Eye (Lond). 2018 Feb;32(2):400-405. doi: 10.1038/eye.2017.201. Epub 2017 Sep 22. PMID 28937146
- [Background] Kinoshita T, Imaizumi H, Miyamoto H, Okushiba U, Hayashi Y, Katome T, Mitamura Y. Changes in metamorphopsia in daily life after successful epiretinal membrane surgery and correlation with M-CHARTS score. Clin Ophthalmol. 2015 Feb 4;9:225-33. doi: 10.2147/OPTH.S76847. eCollection 2015. PMID 25678770
- [Background] Okamoto F, Okamoto Y, Hiraoka T, Oshika T. Effect of vitrectomy for epiretinal membrane on visual function and vision-related quality of life. Am J Ophthalmol. 2009 May;147(5):869-74, 874.e1. doi: 10.1016/j.ajo.2008.11.018. Epub 2009 Feb 6. PMID 19200531
- [Background] McGowan G, Yorston D, Strang NC, Manahilov V. D-CHART: A Novel Method of Measuring Metamorphopsia in Epiretinal Membrane and Macular Hole. Retina. 2016 Apr;36(4):703-8. doi: 10.1097/IAE.0000000000000778. PMID 26441261
- [Background] Klein R, Moss SE, Klein BE, Gutierrez P, Mangione CM. The NEI-VFQ-25 in people with long-term type 1 diabetes mellitus: the Wisconsin Epidemiologic Study of Diabetic Retinopathy. Arch Ophthalmol. 2001 May;119(5):733-40. doi: 10.1001/archopht.119.5.733. PMID 11346401
- [Background] Nichols KK, Mitchell GL, Zadnik K. Performance and repeatability of the NEI-VFQ-25 in patients with dry eye. Cornea. 2002 Aug;21(6):578-83. doi: 10.1097/00003226-200208000-00009. PMID 12131034
- [Background] Orr P, Rentz AM, Margolis MK, Revicki DA, Dolan CM, Colman S, Fine JT, Bressler NM. Validation of the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) in age-related macular degeneration. Invest Ophthalmol Vis Sci. 2011 May 18;52(6):3354-9. doi: 10.1167/iovs.10-5645. PMID 21282568
- [Background] Owen CG, Rudnicka AR, Smeeth L, Evans JR, Wormald RP, Fletcher AE. Is the NEI-VFQ-25 a useful tool in identifying visual impairment in an elderly population? BMC Ophthalmol. 2006 Jun 9;6:24. doi: 10.1186/1471-2415-6-24. PMID 16764714

DOCUMENTS (2):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT04791631/Prot_000.pdf
  • Informed Consent Form (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT04791631/ICF_001.pdf